CLINICAL TRIAL: NCT04508400
Title: Efficacy, Safety and Feasibility of Fosaprepitant for the Prevention of Chemotherapy-induced Nausea and Vomiting in Pediatric Patients With Solid Tumors Receiving Moderately and Highly Emetogenic Chemotherapy
Brief Title: Fosaprepitant for the Prevention of Chemotherapy-induced Nausea and Vomiting in Pediatric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SunYat-senU-fosaprepitant
Record Dates: First submitted 2020-08-09; First posted 2020-08-11 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms | interventions — fosaprepitant; Ondansetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a single dose of fosaprepitant (Experimental): Participants received a single dose of fosaprepitant (age-based adjustment) administered intravenously (IV) on Day 1 prior to chemotherapy plus ondansetron (weight based) IV with dexamethasone (weight based) iv/po prior to chemotherapy and up to 72 hours after chemotherapy.
  Interventions: Drug: Fosaprepitant,ondansetron, dexamethasone
- a single dose of matched placebo (Placebo Comparator): Participants received a single dose of matched placebo for fosaprepitant administered intravenously (IV) on Day 1 prior to chemotherapy plus ondansetron (weight based) IV with dexamethasone (weight based) iv/po prior to chemotherapy and up to 72 hours after chemotherapy.
  Interventions: Drug: placebo ondansetron with dexamethasone

INTERVENTIONS:
Drug: Fosaprepitant,ondansetron, dexamethasone — Participants will randomly assigned 1:1 to receive double-blind study drug ( fosaprepitant plus ondansetron with dexamethasone OR placebo plus ondansetron with dexamethasone). Fosaprepitant or placebo to fosaprepitant were supplied and administered in a blinded manner.
  Other Names: ondansetron, dexamethasone
  Arms: a single dose of fosaprepitant
Drug: placebo ondansetron with dexamethasone — placebo plus ondansetron with dexamethasone
  Other Names: ondansetron, dexamethasone
  Arms: a single dose of matched placebo

SUMMARY:
The purpose is to evaluate the effectiveness and safety of fosaprepitant plus ondansetron with dexamethasone or placebo plus ondansetron with dexamethasone in preventing chemotherapy-induced nausea and vomiting (CINV) with MEC/HE multi-day chemotherapy in children with solid tumors.

DETAILED DESCRIPTION:
Participants will randomly assigned 1:1 to receive double-blind study drug ( fosaprepitant plus ondansetron with dexamethasone OR placebo to fosaprepitant plus ondansetron with dexamethasone). Fosaprepitant or placebo to fosaprepitant were supplied and administered in a blinded manner.

Experimental:

Participants received a single dose of fosaprepitant (age-based adjustment) administered intravenously (IV) on Day 1 prior to chemotherapy plus ondansetron (weight based) IV with dexamethasone (weight based) iv/po prior to chemotherapy and up to 72 hours after chemotherapy.

Placebo Comparator:

Participants received a single dose of matched placebo for fosaprepitant administered intravenously (IV) on Day 1 prior to chemotherapy plus ondansetron (weight based) IV with dexamethasone (weight based) iv/po prior to chemotherapy and up to 72 hours after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Is 6 months to 17 years of age at time of randomization;
2. Participants with solid tumors receiving multi -day chemotherapy associated with moderate or high risk of emetogenicity;
3. Has a preexisting functional central venous catheter available for study drug administration;
4. PS score ≤ 2 points;
5. Has a predicted life expectancy ≥3 months or weight greater than 6Kg;
6. Patient's parent or guardian signs informed consent.

Exclusion Criteria:

1. Has vomited in the 24 hours prior to chemotherapy initiation on Treatment Day 1;
2. Has a symptomatic primary or metastatic central nervous system (CNS) malignancy with nausea and/or vomiting (asymptomatic participants may participate in study);
3. Will be receiving stem cell rescue therapy in conjunction with study-related course of emetogenic chemotherapy or during the 14 days following administration of fosaprepitant/placebo for fosaprepitant;
4. Has received or will receive total body irradiation of radiation therapy to the abdomen or pelvis in the week prior to Treatment Day 1 and/or during the diary reporting period (120 hours following initiation of chemotherapy);
5. Has had benzodiazepine, opioid or opioid like therapy initiated within 48 hours prior to study drug administration, or is expected to receive within 120 hours following initiation of chemotherapy except for single doses of midazolam, temazepam or triazolam;
6. Has started on systemic corticosteroid therapy within 72 hours prior to study drug administration or is expected to receive a corticosteroid as part of the chemotherapy regimen
7. Is currently taking, or has taken within 48 hours of Treatment Day 1 the following drugs with antiemetic properties: 5-hydroxytryptamine 3 (5-HT3) antagonists (e.g., ondansetron), benzamides (e.g., haloperidol), cyclizine, domperidone, herbal therapies with potential antiemetic properties, olanzapine, phenothiazines (e.g., prochlorpenzine), scopolamine (this is not an exhaustive list);
8. Is currently a user of any recreational or illicit drugs (including marijuana) or has current evidence of drug or alcohol abuse or dependence;
9. Is mentally incapacitated or has a significant emotional or psychiatric disorder;
10. Is allergic to fosaprepitant, aprepitant (MK-0869), ondansetron, or any other 5-HT3 antagonist;
11. Has a known history of QT prolongation or is taking any medication that is known to lead to QT prolongation;
12. Has an active infection (e.g., pneumonia), congestive heart failure, bradyarrhythmia, any uncontrolled disease (e.g., diabetic ketoacidosis, gastrointestinal obstruction) except for malignancy;
13. Has ever participated in a previous study of aprepitant or fosaprepitant or has taken an investigational drug with the last 4 weeks;
14. Abnormal liver function (alanine aminotransferase or aspartate aminotransferase ≥ 2 times higher than the upper bound of the normal value) or abnormal renal function (serum creatinine ≥ 2.5 times higher than the upper bound of the normal value);
15. Has participated in a preliminary study of Aprepitant or Fosapretan, or took the study drug in the past 4 weeks;
16. Other situations that the researcher thinks cannot be included.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
CR rate | between 0 and 120 hours after the start of chemotherapy
  Percentage of participants who experienced a complete response (CR; no vomiting/rescue medication) rate in overall phases.

SECONDARY OUTCOMES:
CR rate in acute phase | 0 to 24 Hours Post Initiation of Chemotherapy
  Complete response rate in acute phase
CR rate in delayed phase | 25 to 120 Hours Post Initiation of Chemotherapy
  Complete response rate in delayed phase

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China